CLINICAL TRIAL: NCT00216840
Title: Calcipotriol Plus Betamethasone Dipropionate Gel Compared to Betamethasone Dipropionate in the Gel Vehicle and Calcipotriol in the Gel Vehicle in Scalp Psoriasis
Brief Title: Efficacy and Safety of Calcipotriol Plus Betamethasone Dipropionate Gel in Scalp Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBL 0406 INT
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis of Scalp
MeSH Terms: interventions — calcipotriene; betamethasone-17,21-dipropionate

INTERVENTIONS:
Drug: Calcipotriol plus betamethasone dipropionate (LEO80185 gel)

SUMMARY:
The purpose of the study is to evaluate whether once daily topical treatment for up to 8 weeks of calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate) gel is safe and more effective than betamethasone 0.5 mg/g (as dipropionate) in the gel vehicle and calcipotriol 50 mcg/g in the gel vehicle in patients with scalp psoriasis.

The primary response criterion is the number of patients with absence of disease and very mild disease after 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Scalp psoriasis amenable to topical treatment with a maximum of 100 g of medication per week
* Clinical signs of psoriasis vulgaris on trunk and/or limbs, or earlier diagnosed with psoriasis vulgaris on trunk and/or limbs
* Extent of scalp psoriasis involving more than 10% of the total scalp area
* Investigator's assessment of clinical signs of the scalp of at least 2 in one of the clinical signs, erythema, thickness and scaliness, and at least 1 in each of the other two clinical signs
* Disease severity on the scalp graded as Mild, Moderate, Severe or Very severe according to the investigator's global assessment of disease severity

Exclusion Criteria:

* PUVA or Grenz ray therapy within 4 weeks prior to randomisation
* UVB therapy within 2 weeks prior to randomisation
* Systemic treatment with biological therapies, with a possible effect on scalp psoriasis within 6 months prior to randomisation
* Systemic treatment with all other therapies than biologicals, with a possible effect on scalp psoriasis (e.g., corticosteroids, vitamin D analogues, retinoids, immunosuppressants) within 4 weeks prior to randomisation
* Any topical treatment of the scalp (except for medicated shampoos and emollients) within 2 weeks prior to randomisation
* Topical treatment of the face, trunk and/or limbs with very potent WHO group IV corticosteroids within 2 weeks prior to randomisation
* Current diagnosis of erythrodermic, exfoliative or pustular psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350
Dates: Start 2004-12; Study Completion 2005-09

PRIMARY OUTCOMES:
- Patients with "Controlled disease" ("Absence of disease" or "Very mild disease") according to investigator's global assessment of disease severity at week 8.

SECONDARY OUTCOMES:
- Total sign score at week 8
- Score for scaliness, redness and thickness at week 8
- Patients with "Controlled disease" ("Absence of disease" or "Very mild disease") according to investigator's global assessment of disease severity at week 2 and 4
- Patients with "Treatment success" ("Almost clear" or "Cleared") according to patient's overall assessment of disease severity at week 8
- Evaluation of Adverse Events
- Evaluation of Laboratory Data

CONTACTS AND LOCATIONS:
Overall Officials: Peter van de Kerkhof, MD, Principal Investigator — Universitair Medisch, Afdeling Dermatologie
Locations (7):
- Universitair Ziekenhuis Sint Rafaël, Dienst Dermatologie, Leuven, Belgium
- Innovaderm Research Inc., Montreal, Quebec, Canada
- Policlinic of Dermatology, Medical Reception Centre, Turku, Finland
- Hôpital Trousseau, Service de Dermatologie CHU Tours, Tours, France
- Georg-August-Universität Göttingen, Abteilung Dermatologie und Venerologie, Göttingen, Germany
- Universitair Medisch, Centrum St. Radboud, Afdeling Dermatologie, Nijmegen, Netherlands
- Royal Gwent Hospital, Department of Dermatology, Newport, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van de Kerkhof PC, Hoffmann V, Anstey A, Barnes L, Bolduc C, Reich K, Saari S, Segaert S, Vaillant L. A new scalp formulation of calcipotriol plus betamethasone dipropionate compared with each of its active ingredients in the same vehicle for the treatment of scalp psoriasis: a randomized, double-blind, controlled trial. Br J Dermatol. 2009 Jan;160(1):170-6. doi: 10.1111/j.1365-2133.2008.08927.x. Epub 2008 Nov 25. PMID 19067709
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en